CLINICAL TRIAL: NCT06438848
Title: Effects of a Physical Therapy Program Combined With Manual Lymphatic Drainage on Shoulder Function, , and Pain in Breast Cancer Patients With Axillary Web Syndrome Following Axillary Dissection: A Randomized Controlled Trial
Brief Title: Effects of Lymph Drainage on Patients With Axillary Web Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taif University (Other)
Responsible Party: Principal Investigator, Ibrahim Mohammad Alkayshan, Physical therapist, Taif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-1241
Record Dates: First submitted 2024-05-22; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Intervention Model Description: Controlled parallel groups
Who Masked: Participant, Care Provider
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy program (Experimental): group will be prescribed a usual physical therapy program three times a week for four weeks, which will be conducted in the clinic. The program consists of eight sessions comprising warm-up and cool-down, stretching activities, and strengthening exercises, and manual therapy. The program will start with 10-minute warm-up and 10-minute cool-down periods of physical therapy sessions
  Interventions: Other: Physical therapy program
- Physical therapy program with lymphedema drainage (Experimental): physical therapy program three times a week for four weeks, which will be conducted in the clinic. The program consists of eight sessions comprising warm-up and cool-down, stretching activities, and strengthening exercises,And manual lymphatic drainage prescribed 20 minutes of MLD daily. The program will be prescribed five times a week, for four weeks
  Interventions: Other: Physical therapy program with lymphedema drainage

INTERVENTIONS:
Other: Physical therapy program — group will be prescribed a usual physical therapy program three times a week for four weeks, which will be conducted in the clinic. The program consists of eight sessions comprising warm-up and cool-down, stretching activities, and strengthening exercises, and manual therapy. The program will start with 10-minute warm-up and 10-minute cool-down periods of physical therapy sessions
  Arms: Physical therapy program
Other: Physical therapy program with lymphedema drainage — physical therapy program three times a week for four weeks, which will be conducted in the clinic. The program consists of eight sessions comprising warm-up and cool-down, stretching activities, and strengthening exercises,And manual lymphatic drainage prescribed 20 minutes of MLD daily. The program will be prescribed five times a week, for four weeks
  Arms: Physical therapy program with lymphedema drainage

SUMMARY:
Effects of a physical therapy program combined with manual lymphatic drainage on shoulder pain and function, quality of life, lymphedema incidence in breast cancer patients with axillary web syndrome following axillary dissection: A randomized controlled trial.

DETAILED DESCRIPTION:
This study's objective is to assess the effectiveness of physical therapy (PT) combined with manual lymphatic drainage (MLD) on shoulder pain and function, lymphedema, visible cords, and quality of life (QOL), compared to physical therapy alone, in subjects with breast cancer and suffering of axillary web syndrome (AWS).

ELIGIBILITY:
Inclusion Criteria:

* had a breast cancer dissection with lymphadenectomy and/or sentinel lymph node biopsy and a subsequent appearance of AWS (diagnosed by physical examination and also by using the Screening Test AWS (ST-AWS)) [35].

  * suffering of pain that exceeds 6-8 points (measured by the numeric rating scale (NRS)) in the region of the cording on the upper/lower arm, elbow, and dorsum site, and
  * have visible or palpable cords in the arm or breast.

Exclusion Criteria:

* suffering of both acute thrombosis and lymphedema,

  * suffering of skin issues like infections or musculoskeletal conditions like adhesive capsulitis, rheumatoid arthritis, pectoral muscle tightness, and diseases of the rotator cuff, and/or
  * having cording that doesn't involve an arm and only affects the chest or side of the thorax.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 5 weeks
  Pain intensity will be assessed using the NRS (0-10). A score of 0 means there is no pain, while a score of 10 means presence of severe pain.
Disability | 5 weeks
  Assessment of disability will be done using the Arabic Quick-DASH questionnaire which is an 11-item self-report questionnaire, The DASH has five response options for each item from 0=no difficulty to perform or no symptoms to 5=unable to do. A higher score reflects greater disability.

SECONDARY OUTCOMES:
Limb Girth | 4 weeks
  The limb girth will be measured using the tape measurement. Upper limb volumes will be calculated from circumference measurements taken at 4-cm intervals from the dorsum of the wrist to the axilla. The diagnostic criterion for lymphedema was ≥3 % volume increase from baseline in the affected upper limb.
Cording | 5 weeks
  lymphedema therapist (PT/CLT) will examine the arm and axilla for any visible or palpable cords. The findings will be either positive for cording or negative. It is a nominal qualitative variable.
Muscular strength | 5 weeks
  Using a hand-held dynamometer, the maximum voluntary isometric contraction of the muscles will be used to assess their strength.
Range of motion | 5 weeks
  The active ROM (AROM) will be assessed using a goniometer which has been proved to have reliability and concurrent validity for measuring shoulder mobility measurements
Quality of life for participants | 5 weeks
  The EORTC QLQ-C30 is a 30-item questionnaire including measuring Global Health status (2 items), Functional scales (15 items) and Symptoms scales/items (13 items). Items were measured using a 4-point Likert Scale ranging from Not at all (1) to Very much (4)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Alzahrani, PHD, Study Chair — Taif University

IPD SHARING:
Plan to Share IPD: No